CLINICAL TRIAL: NCT03942497
Title: Clinical-pathological Characterization and Outcomes of Metastatic Urothelial Cancer in Latin America: Retrospective and Translational Multicenter Database
Brief Title: Clinical-pathological Characterization and Outcomes of Metastatic Urothelial Cancer in Latin America
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 1518
Record Dates: First submitted 2019-04-25; First posted 2019-05-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2022-09

CONDITIONS: Recurrent/Metastatic Urothelial Cancers
Keywords: metastatic; recurrent; urothelial cancers; renal pelvis; ureter; bladder; urethra
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Archived tumor samples from Formalin-Fixed Paraffin-Embedded (FFPE) blocks or slides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The LACOG 1518 study will characterize demographic and clinical-pathological profile of patients diagnosed with recurrent/ metastatic urothelial cancer in Latin America.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years;
2. Histological confirmation of urothelial carcinoma (include mixed urothelial histology);
3. Diagnosis of recurrent or metastatic (Stage IV) urothelial carcinoma during the period of January 2016 to July 2018;
4. Site and investigator ability to collect adequate patient characteristics, treatment and outcome data from medical records;
5. Availability of tumor sample (FFPE/slides) from primary tumor or metastatic site at the time of registration.

Exclusion Criteria:

1. Synchronous tumors or history of other malignancy in the previous 3 years before study entry (exception to non-melanoma skin cancer or non-invasive cancers);
2. Pure non-urothelial carcinoma histology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent/ metastatic urothelial carcinoma diagnosed between January 2016 to July 2018.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Epidemiology | 2 years
  Overall survival (OS) will be defined from the date of treatment initiation to date of death from any cause. In case of patients that received palliative care only, OS will be defined from date of diagnosis of advanced disease to date of death from any cause. Patients who are alive will be censored at the date of last known contact.

SECONDARY OUTCOMES:
Socioeconomic chactacteristcs | 2 years
  Health Care Insurance (Public or Private)
Overall response | 2 years
  Defined as the proportion of patients who have a partial or complete response to therapy according to RECIST 1.1
Duration of response | 2 years
  Defined as the time from response to progression by RECIST v11.1 or death
PFS | 2 years
  Progression-free survival (PFS) will be defined from date of treatment initiation to date of disease progression or death from any cause, whichever occurs first in each line.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (9):
- Brazil (9):
  - CLION, Salvador, Estado de Bahia
  - Clínica AMO, Salvador, Estado de Bahia
  - Hospital São Rafael, Salvador, Estado de Bahia
  - LIGA, Curitiba, Paraná
  - CPO Pucrs, Porto Alegre, Rio Grande do Sul
  - CEPON, Florianópolis, Santa Catarina
  - Beneficência Portuguesa, São Paulo, São Paulo
  - Centro Paulista de Oncologia, São Paulo, São Paulo
  - Sírio Libanês, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Milowsky MI, Rumble RB, Booth CM, et al. Guideline on Muscle-Invasive and Metastatic Bladder Cancer (European Association of Urology Guideline): American Society of Clinical Oncology Clinical Practice Guideline Endorsement. J Clin Oncol. 2016;34(16):1945-1952. doi:10.1200/JCO.2015.65.9797 2. Instituto Nacional de Câncer José Alencar Gomes. Estimativa 2018: Incidência de Câncer No Brasil. Rio de Janeiro: INCA; 2018. http://www.inca.gov.br/estimativa/2018. 3. International Agency for Research on Cancer, International Association of Cancer Registries. Cancer Incidence in Five Continents. Volume X Volume X.; 2014. http://www.iarc.fr/en/publications/pdfs-online/epi/sp164/. Accessed November 21, 2018. 4. Secretaria de Estado da Saúde de São Paulo. FOSP - Fundação Oncocentro de São Paulo. http://www.fosp.saude.sp.gov.br/. Accessed October 30, 2018. 5. Edwards IR, Aronson JK. Adverse drug reactions: definitions, diagnosis, and management. Lancet. 2000;356(9237):1255-1259. doi:10.1016/S0140-6736(00)02799-9